CLINICAL TRIAL: NCT02311868
Title: Effect of Short-term Synbiotic Treatment on Plasma P-cresol Levels in Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-cres Probinul
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Hemodialysis
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SYNBIOTIC (Experimental): Patients of this group assumed Probinul-Neutro® po 5g three times a day for 30 day
  Interventions: Dietary Supplement: SYNBIOTIC (Probinul neutro®)
- Placebo (Placebo Comparator): patients of this group received 5g of placebo 3 times a day for 30 days
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: SYNBIOTIC (Probinul neutro®) — Probinul neutro® assumed three times a day far from meals as 5 g powder packets dissolved in water. Probinul neutro® contains 5×109 Lactobacillus plantarum, 2×109 Lactobacillus casei subp. rhamnosus and 2×109 Lactobacillus gasseri, 1×109 Bifidobacterium infantis and 1×109 Bifidobacterium longum, 1×109 Lactobacillus acidophilus, 1×109 Lactobacillus salivarus and 1×109 Lactobacillus sporogenes and 5×109 Streptococcus termophilus, prebiotic inulin (2.2 g; VB Beneo Synergy 1) and 1.3 g of tapioca-resistant starch.
  Other Names: PROBINUL
  Arms: SYNBIOTIC
Dietary Supplement: PLACEBO — Tapioca-resistant starch powder similar in colour, texture and taste to the symbiotic mixture, assumed three times a day far from meals as 5 g powder packets dissolved in water.
  Arms: Placebo

SUMMARY:
The interest on gastrointestinal (GI) dysfunction in hemodialysis has been growing in the last years. it is now accepted that GI dysfunction in dialyzed patients may contribute to systemic microinflammation by promoting gut dysbiosis and bacterial translocation in the blood. Another mechanism by which GI dysfunction contributes to systemic symptoms is related to metabolic activity of the dysbiotic microflora growing in the gut of these patients to generate toxic compounds such as phenols, indoles, and amines. Epidemiological evidence has strongly linked one of these compounds, p-Cresol, to cardiovascular risk and mortality in hemodialysis patients. In the present paper the investigators investigated the effect of a probiotic/prebiotic mixture on plasma p-cresol concentrations and GI symptoms and in hemodialysis patients.

DETAILED DESCRIPTION:
In patients with end stage renal disease, alterations in gut microbioma are posited to be responsible for gastrointestinal symptoms and generation of p-cresol, a uremic toxin, that has been associated to cardiovascular mortality.

This double blind randomized placebo controlled pilot study evaluates whether Probinul-neutro®, a synbiotic preparation that normalizes intestinal microflora, may lower plasma p-cresol concentrations and reduce gastrointestinal symptoms in hemodialysis patients.

Thirty patients on hemodialysis were randomized to receive either Probinul neutro® or placebo for four weeks. Total plasma p-cresol concentrations was assessed at baseline, and 15 and 30 days after treatment start. At the same study times, ease and frequency of defecation, upper and lower abdominal pain, stool shape, borborygmi and flatus were quantified by subjective assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis
* age >18 years

Exclusion Criteria:

* severe infections
* diabetes
* malignancy
* history of food intolerance
* autoimmune disorders
* severe malnutrition
* clinical conditions requiring artificial feeding
* kidney transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma p-cresol concentration | 30 days
  Fasting blood samples were drawn for the p-cresol plasma level

SECONDARY OUTCOMES:
composite outcome of gastrointestinal symptoms | 30 days
  Patients were asked to fill in a form for the scored evaluation of gastrointestinal symptoms (upper and inferior abdominal pain, borborygmus and flatus defecation frequency or easeand stool), and stool shape (Bristol stool chart)

CONTACTS AND LOCATIONS:
Locations (1):
- federico II university, department of nephrology, Naples, Italy, Italy